CLINICAL TRIAL: NCT00398086
Title: A Phase I Trial of Gemcitabine (Gemzar) Plus ABI-007 (ABRAXANE) In Patients With Advanced Metastatic Pancreatic Cancer
Brief Title: Gemcitabine Plus Albumin-bound Paclitaxel In Patients With Advanced Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA040
Record Dates: First submitted 2006-11-08; First posted 2006-11-10 (Estimated); Results first posted 2013-08-21 (Estimated); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: Metastatic Pancreatic Cancer, Abraxane, Gemcitabine
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 100 mg/m^2 (Experimental): Participants received albumin-bound paclitaxel 100 mg/m^2 followed by gemcitabine 1000 mg/m^2 by intravenous infusion (IV) on Days 1, 8 and 15 of each 28 day cycle (dose level one). Treatment continued until progressive disease or unacceptable toxicity.
  Interventions: Drug: Gemcitabine; Drug: Albumin-bound paclitaxel
- 125 mg/m^2 (Experimental): Participants received albumin-bound paclitaxel 125 mg/m^2 followed by gemcitabine 1000 mg/m^2 by intravenous infusion (IV) on Days 1, 8 and 15 of each 28 day cycle (dose level two). Treatment continued until progressive disease or unacceptable toxicity.
  Interventions: Drug: Gemcitabine; Drug: Albumin-bound paclitaxel
- 150 mg/m^2 (Experimental): Participants received albumin-bound paclitaxel 150 mg/m^2 followed by gemcitabine 1000 mg/m^2 by intravenous infusion (IV) on Days 1, 8 and 15 of each 28 day cycle (dose level three). Treatment continued until progressive disease or unacceptable toxicity.
  Interventions: Drug: Gemcitabine; Drug: Albumin-bound paclitaxel

INTERVENTIONS:
Drug: Gemcitabine — Administered by intravenous infusion over 30 minutes.
  Other Names: Gemzar®
Drug: Albumin-bound paclitaxel — Administered by intravenous infusion over 30 minutes.
  Other Names: ABI-007; ABRAXANE®

SUMMARY:
To determine the maximum tolerated dose and dose-limiting toxicity of Gemcitabine plus Albumin-bound paclitaxel (ABI-007) in patients with advanced metastatic pancreatic cancer.

DETAILED DESCRIPTION:
Albumin-bound paclitaxel is a novel, solvent-free, albumin-bound, 130 nanometer particle form of paclitaxel designed to avoid the problems associated with solvents used in Taxol(Abraxane prescribing information 2005). Albumin has a number of properties that make it an attractive molecule to combine with paclitaxel. Albumin is a natural transporter of endogenous hydrophobic molecules such as water-insoluble vitamins and hormones (Vorum 1999)and albumin binding to the gp-60 receptor (albondin) initiates the caveolae-mediated endothelial transport of protein-bound and unbound plasma constituents (John et al 2003, Minshall et al 2003, Tiruppathi et al 1997).

This study consisted of a Phase 1 dose escalation phase, a Phase 2 treatment phase and a 24-month follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

* Patient has histologically or cytologically confirmed metastatic adenocarcinoma of the pancreas. Patients with islet cell neoplasms are excluded.
* Male or non-pregnant and non-lactating female, and age greater or equal to 18.

  * If a female patient is of child-bearing potential, as evidenced by regular menstrual periods, she must have a negative serum pregnancy test beta-human chorionic gonadotropin (B-hCG) documented within 72 hours of the first administration of study drug.
  * If sexually active, the patient must agree to use contraception considered adequate and appropriate by the investigator.
* Patient must have received no prior therapy for the treatment of metastatic disease. Prior treatment with 5-fluorouracil (5-FU) or gemcitabine administered as a radiation sensitizer during and up to 4 weeks after radiation therapy is allowed. If a patient received gemcitabine in the adjuvant setting, tumor recurrence must have occurred at least 6 months after completing the last dose of gemcitabine.
* Patient has the following blood counts at baseline

  * Absolute neutrophil count (ANC) equal or greater to 1.5 x 10^9/L;
  * Platelets equal or greater to 100 x 10^9/L
  * Hemoglobin equal or greater to 9 g/dL.
  * Patient has the following blood chemistry levels at baseline:
  * Aspartate aminotransferase (SGOT), Alanine aminotransferase (SGPT) equal or less than 2.5 x upper limit of normal range (ULN) is allowed
  * Bilirubin less than or equal to ULN
  * Serum creatinine within normal limits or calculated clearance equal or greater to 60 mL/min/1.73M^2 patients with serum creatinine levels above the institutional normal value
* Patient has no clinically significant abnormalities in urinalysis results
* Patient has acceptable coagulation status as indicated by a prothrombin time (PT) within normal limits (plus or minus 15%) and partial thromboplastin time (PTT) within normal limits (plus or minus 15%).
* Patient has a Karnofsky performance status (KPS) greater or equal to 70 (Eastern Cooperative Oncology Group [ECOG] PS 0-1).
* Patient has one or more metastatic tumors measurable by computed tomography (CT) scan.
* Patient has been informed about the nature of study, and has agreed to participate in the study, and signed the Informed Consent form prior to participation in any study-related activities.

Exclusion Criteria:

* Patient has known brain metastases unless previously treated and well controlled for at least 3 months (defined as stable clinically, no edema, no steroids and stable in two scans at least 4 weeks apart).
* Patient uses therapeutic coumadin for a history of pulmonary emboli and deep vein thrombosis (DVT).
* Patient has active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy.
* Patient has known infection with human immunodeficiency virus (HIV), hepatitis B, hepatitis C.
* Patient has undergone major surgery, other than diagnostic surgery i.e.-- done to obtain a biopsy for diagnosis without removal of an organ), with 4 weeks prior to Day 1 of treatment in this study.
* Patient received radiotherapy, surgery, chemotherapy, or an investigational therapy within 3 weeks prior to study entry weeks (6 weeks for nitrosureas or mitomycin C).
* Patient has a history of allergy or hypersensitivity to the study drug.
* Patient has serious medical risk factors involving any of the major organ systems such that the investigator considers it unsafe for the patient to receive an experimental research drug.
* Patient is unwilling or unable to comply with study procedures.
* Patient is enrolled in any other clinical protocol or investigational trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2006-11-01 (Actual); Primary Completion 2008-09-01 (Actual); Study Completion 2010-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Von Hoff, MD, Principal Investigator — Scottsdale Clinical Research Institute
Locations (5):
- United States (5):
  - University of Alabama at Birmingham Comprehensive Cancer Ctr, Birmingham, Alabama
  - Scottsdale Healthcare/Virginia Pipe Cancer Institute, Scottsdale, Arizona
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins University, Baltimore, Maryland
  - Virigina Piper Cancer Institute, Minneapolis, Minnesota
  - South Texas Oncology & Hematology, San Antonio, Texas

REFERENCES:
- [Background] Von Hoff DD, Ramanathan RK, Borad MJ, Laheru DA, Smith LS, Wood TE, Korn RL, Desai N, Trieu V, Iglesias JL, Zhang H, Soon-Shiong P, Shi T, Rajeshkumar NV, Maitra A, Hidalgo M. Gemcitabine plus nab-paclitaxel is an active regimen in patients with advanced pancreatic cancer: a phase I/II trial. J Clin Oncol. 2011 Dec 1;29(34):4548-54. doi: 10.1200/JCO.2011.36.5742. Epub 2011 Oct 3. PMID 21969517
- [Derived] Korn RL, Von Hoff DD, Borad MJ, Renschler MF, McGovern D, Curtis Bay R, Ramanathan RK. 18F-FDG PET/CT response in a phase 1/2 trial of nab-paclitaxel plus gemcitabine for advanced pancreatic cancer. Cancer Imaging. 2017 Aug 3;17(1):23. doi: 10.1186/s40644-017-0125-5. PMID 28774338

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was initiated in November 2006 and completed in September 2008. Sixty-seven patients were enrolled at four sites in the US.
Pre-assignment Details: In Phase 1, patients were assigned sequentially to one of the three potential dose levels based on the dose cohort currently enrolling patients (a total of 30 patients). After the maximum tolerated dose (MTD) was determined, all subsequent patients were enrolled at that dose level in Phase 2 (37 patients).
Period: Overall Study
Arm/Group | 100 mg/m^2 | 125 mg/m^2 | 150 mg/m^2
Started | 20 | 44 | 3
Phase 1, Dose Escalation Population | 20 | 7 | 3
Completed | 11 (Completed defined as discontinuation due to progressive disease.) | 21 (Completed defined as discontinuation due to progressive disease.) | 1 (Completed defined as discontinuation due to progressive disease.)
Not Completed | 9 | 23 | 2
Not completed — Unacceptable Toxicity | 2 | 8 | 2
Not completed — Adverse Event | 1 | 4 | 0
Not completed — Physician Decision | 1 | 4 | 0
Not completed — Withdrawal by Subject | 5 | 7 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 100 mg/m^2 | 125 mg/m^2 | 150 mg/m^2 | Total
Number analyzed (Participants) | 20 | 44 | 3 | 67
Age, Continuous [Median (Full Range); unit: years] | 62.0 [30 to 86] | 61.5 [28 to 78] | 69.0 [53 to 72] | 62.0 [28 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 25 | 1 | 35
  Male | 11 | 19 | 2 | 32
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 1 | 0 | 2
  Black, of African Heritage | 0 | 2 | 0 | 2
  White, Non-Hispanic, and Non-Latino | 16 | 37 | 1 | 54
  White, Hispanic, or Latino | 2 | 4 | 2 | 8
  Other | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 20 | 44 | 3 | 67
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — A scale used to assess the progress of disease in a patient, how the disease affects the daily living abilities of the patient, and determine appropriate treatment and prognosis.
  participants
    0 (Fully Active) | 9 | 22 | 2 | 33
    1 (Restrictive but Ambulatory) | 11 | 22 | 1 | 34
Histology of Primary Diagnosis: Adenocarcinoma [Number; unit: participants] | 20 | 44 | 3 | 67
Time from First Documented Metastasis/Relapse to Study Entry [Median (Full Range); unit: months] | 0.8 [0 to 11] | 0.7 [0 to 13] | 0.3 [0 to 1] | 0.7 [0 to 13]
Current Site(s) of Metastasis/Relapse [Number; unit: participants] — Patients could be in multiple sites of metastasis/relapse categories.
  participants
    Skin/Soft Tissue | 0 | 1 | 0 | 1
    Supraclavicular Nodes | 0 | 2 | 0 | 2
    Axilla | 2 | 0 | 0 | 2
    Bone | 1 | 3 | 0 | 4
    Lung/Thoracic | 5 | 18 | 1 | 24
    Liver | 11 | 33 | 2 | 46
    Abdomen/Peritoneum | 16 | 37 | 1 | 54
    Pelvis | 1 | 3 | 1 | 5
    Other | 8 | 6 | 0 | 14
Dominant Current Site of Metastasis/Relapse [Number; unit: participants]
  Visceral | 19 | 44 | 3 | 66
  Non-visceral | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities
Description: A dose-limiting toxicity (DLT) is defined as one or more of the following toxicities related to study drug during Cycle 1, according to the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE), Version 3:
  * Grade 4 neutropenia lasting >3 days in the absence of growth factor support;
  * Grade 4 neutropenia associated with fever >38.5°C;
  * Any other Grade 4 hematological toxicity;
  * Grade 3 thrombocytopenia with hemorrhage;
  * Grade 3 or 4 nausea, vomiting or diarrhea despite prophylaxis or treatment with an optimal anti-emetic or anti-diarrhea regimen;
  * Any other Grade 3 or higher non-hematological toxicity attributable to the study drug, excluding alopecia and fatigue.
Time Frame: Cycle 1 (Days 1-28)
Population: Phase 1 treated population
Measure: Number; unit: participants
Arm/Group | 100 mg/m^2 | 125 mg/m^2 | 150 mg/m^2
Number analyzed (Participants) | 20 | 7 | 3
participants | 4 | 0 | 1

2. Secondary Outcome: Number of Participants With Adverse Events (AE)
Description: An AE was any untoward medical occurrence, not necessarily having a causal relationship with the patient's treatment, that began or worsened in grade after the start of study drug through 30 days after the last dose.
  A serious AE (SAE) is any untoward medical occurrence that is fatal, life-threatening, results in persistent or significant disability or incapacity, requires or prolongs existing in-patient hospitalization, is a congenital anomaly/birth defect, or is a condition that may jeopardize the patient or may require intervention to prevent one of the outcomes listed above.
  Treatment-related AEs (TRAEs) include those assessed by the Investigator as possibly, probably, or definitely related to study treatment.
  Severity was graded according to the NCI CTCAE based on the following: Grade 1- Mild; Grade 2 -Moderate; Grade 3 - Severe; Grade 4 - Life-threatening or disabling; Grade 5 - Death related to AE.
Time Frame: Up to 25 months
Population: Treated patients: all enrolled patients who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | 100 mg/m^2 | 125 mg/m^2 | 150 mg/m^2
Number analyzed (Participants) | 20 | 44 | 3
participants
  Patients with at least 1 AE | 20 | 44 | 3
  At least 1 grade 3 or higher AE | 15 | 42 | 3
  At least 1 treatment-related AE | 18 | 42 | 3
  At least 1 treatment-related grade 3 to 5 AE | 11 | 38 | 3
  Patients with at least 1 SAE | 10 | 24 | 1
  Patients with at least 1 treatment-related SAE | 4 | 12 | 1
  At least 1 AE and drug permanently discontinued | 3 | 12 | 2
  At least 1 TRAE and drug permanently discontinued | 2 | 8 | 2
  At least 1 dose reduction due to TRAE | 4 | 10 | 1
  At least 1 dose interruption due to AE | 1 | 0 | 0
  At least 1 treatment-related AE dose interruption | 1 | 0 | 0
  At least 1 treatment-emergent dose delay due to AE | 14 | 27 | 3
  At least 1 treatment-related dose delay due to AE | 13 | 27 | 3
  At least 1 AE resulting in death | 0 | 1 | 1

3. Secondary Outcome: Percentage of Participants Who Achieved an Objective Confirmed Overall Response
Description: Overall Response is defined as the percent of participants who achieve an objective confirmed complete (CR) or partial response (PR). Response was determined according to Response Evaluation Criteria in Solid Tumors (RECIST) guidelines, assessed by an Independent Radiological Reviewer.
  CR: The disappearance of all known disease and no new sites or disease-related symptoms confirmed at least 4 weeks after initial documentation. All sites must be assessed, including non-measurable sites, such as effusions, or markers.
  PR: At least a 30% decrease in the sum of the longest diameters of target lesions, taking as a reference the baseline sum of the longest diameters confirmed at least 4 weeks after initial documentation and no new non-target lesions and/or unequivocal progression of existing non-target lesions. PR is also recorded when all measurable disease has completely disappeared, but a non-measurable component (i.e., ascites) is still present but not progressing.
Time Frame: Up to approximately 4 years
Population: Treated patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 100 mg/m^2 | 125 mg/m^2 | 150 mg/m^2
Number analyzed (Participants) | 20 | 44 | 3
percentage of participants | 25 [8.7 to 49.1] | 39 [24.2 to 53.0] | 0 [NA to NA] — Could not be calculated as no participants responded in this group

4. Secondary Outcome: Percentage of Participants With Disease Control
Description: Disease control is defined as participants with Stable Disease for at least 16 weeks, or confirmed complete or partial overall response, based on RECIST guidelines and assessed by an Independent Radiological Reviewer.
  Stable disease is defined as neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for Progressive Disease, and no new non-target lesions or unequivocal progression of existing non-target lesions. Progressive Disease is defined as at least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum of the longest diameters recorded since the treatment started; or the appearance of one or more new lesions; or the unequivocal progression of a non-target lesion.
Time Frame: Up to approximately 4 years
Population: Treated patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 100 mg/m^2 | 125 mg/m^2 | 150 mg/m^2
Number analyzed (Participants) | 20 | 44 | 3
percentage of participants | 55 [33.2 to 76.8] | 55 [39.8 to 69.3] | 33 [0.8 to 90.6]

5. Secondary Outcome: Progression-free Survival
Description: Progression-free survival is defined as the time from first dose of study drug to the start of disease progression or patient death, whichever occurs first, assessed by an Independent Radiological Reviewer. Participants who do not have disease progression or have not died were censored at the last known time that the participant was progression free. Progression-free survival was summarized using Kaplan-Meier methods.
  Progressive Disease is defined as at least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum of the longest diameters recorded since the treatment started; or the appearance of one or more new lesions; or the unequivocal progression of a non-target lesion.
Time Frame: Up to approximately 4 years
Population: Treated patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 100 mg/m^2 | 125 mg/m^2 | 150 mg/m^2
Number analyzed (Participants) | 20 | 44 | 3
months | 6.1 [3.7 to NA] — Could not be estimated due to low number of events. | 6.9 [4.8 to 9.2] | 1.6 [0.5 to 10.0]

6. Secondary Outcome: Duration of Response
Description: Duration of response was assessed by progression-free survival for participants who achieved a confirmed Complete Response or Partial Response, assessed by an Independent Radiological Reviewer.
Time Frame: Up to approximately 4 years
Population: Treated patients with an overall confirmed Complete Response or Partial Response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 100 mg/m^2 | 125 mg/m^2 | 150 mg/m^2
Number analyzed (Participants) | 5 | 17 | 0
months | NA [2.4 to NA] — Not estimable due to the low number of events. | 7.3 [5.5 to 21.9] |

7. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from the date of first dose of study drug to the date of patient death from all causes. Participants who did not die were censored at the last known time the patient was alive. Patient survival was summarized using Kaplan-Meier methods.
Time Frame: Up to approximately 4 years
Population: Treated patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 100 mg/m^2 | 125 mg/m^2 | 150 mg/m^2
Number analyzed (Participants) | 20 | 44 | 3
months | 9.3 [6.6 to 11.9] | 12.2 [8.9 to 17.9] | 6.1 [0.5 to 17.9]

8. Secondary Outcome: Maximal Degree of Myelosuppression
Description: The maximal degree of myelosuppression was assessed by the overall nadir of absolute neutrophil count (ANC), white blood cell count and platelet count based on clinical laboratory measurements.
Time Frame: During the treatment phase, up to a maximum of 24 months.
Population: Treated patients with available data
Measure: Mean (Standard Deviation); unit: x10^9/L
Arm/Group | 100 mg/m^2 | 125 mg/m^2 | 150 mg/m^2
Number analyzed (Participants) | 20 | 43 | 3
x10^9/L
  Absolute neutrophil count | 1.38 (1.541) | 0.96 (1.446) | 0.47 (0.460)
  White blood cell count | 2.69 (1.734) | 2.18 (1.849) | 1.52 (1.484)
  Platelet count | 120.3 (79.02) | 88.3 (62.10) | 58.7 (48.64)

9. Secondary Outcome: Maximal Degree of Anemia
Description: The maximal degree of anemia (and myelosuppression) was assessed by the overall (any time after first dose of study drug) nadir of hemoglobin levels based on clinical laboratory measurements.
Time Frame: During the treatment phase, up to a maximum of 24 months.
Population: Treated patients with available data
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | 100 mg/m^2 | 125 mg/m^2 | 150 mg/m^2
Number analyzed (Participants) | 20 | 43 | 3
g/L | 95.1 (12.85) | 91.8 (10.43) | 95.3 (15.37)

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to 30 days after the last dose (a maximum of 25 months).
Arm/Group | 100 mg/m^2 | 125 mg/m^2 | 150 mg/m^2
Serious Adverse Events (participants affected / at risk) | 10/20 | 24/44 | 1/3
Other Adverse Events (participants affected / at risk) | 20/20 | 44/44 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 100 mg/m^2 (N=20) | 125 mg/m^2 (N=44) | 150 mg/m^2 (N=3)
Pneumonia (Infections and infestations) | 1 | 2 | 0
Bacteraemia (Infections and infestations) | 0 | 2 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 1 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0
Endocarditis (Infections and infestations) | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 2 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Duodenal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Enterocutaneous fistula (Gastrointestinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Obstruction gastric (Gastrointestinal disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 3 | 0
Pain (General disorders) | 2 | 0 | 0
Hernia obstructive (General disorders) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 0
Migraine with aura (Nervous system disorders) | 0 | 1 | 0
Sedation (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 3 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Medical device complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0
Ureteric obstruction (Renal and urinary disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 100 mg/m^2 (N=20) | 125 mg/m^2 (N=44) | 150 mg/m^2 (N=3)
Anaemia (Blood and lymphatic system disorders) | 12 | 30 | 2
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 4 | 18 | 2
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 10 | 25 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 26 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 1 | 1 | 0
Tachycardia (Cardiac disorders) | 2 | 2 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 2 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 0
Steroid withdrawal syndrome (Endocrine disorders) | 1 | 0 | 0
Blepharitis (Eye disorders) | 1 | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 1 | 0 | 0
Diplopia (Eye disorders) | 1 | 0 | 0
Dry eye (Eye disorders) | 1 | 1 | 0
Eye swelling (Eye disorders) | 1 | 1 | 0
Vision blurred (Eye disorders) | 2 | 2 | 0
Visual impairment (Eye disorders) | 1 | 3 | 0
Abdominal distension (Gastrointestinal disorders) | 4 | 9 | 1
Abdominal pain (Gastrointestinal disorders) | 7 | 17 | 2
Abdominal pain lower (Gastrointestinal disorders) | 3 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 4 | 0
Colitis (Gastrointestinal disorders) | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 6 | 21 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 23 | 2
Dry mouth (Gastrointestinal disorders) | 3 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 5 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 1 | 0
Eructation (Gastrointestinal disorders) | 1 | 1 | 0
Faecal incontinence (Gastrointestinal disorders) | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 2 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 3 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 3 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 3 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 2 | 1
Nausea (Gastrointestinal disorders) | 8 | 29 | 2
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 0
Oral mucosal erythema (Gastrointestinal disorders) | 1 | 1 | 0
Oral pain (Gastrointestinal disorders) | 2 | 1 | 0
Retching (Gastrointestinal disorders) | 1 | 2 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 1 | 0
Vomiting (Gastrointestinal disorders) | 5 | 20 | 2
Asthenia (General disorders) | 1 | 7 | 1
Catheter related complication (General disorders) | 1 | 0 | 0
Catheter site inflammation (General disorders) | 1 | 0 | 0
Chest discomfort (General disorders) | 2 | 1 | 0
Chest pain (General disorders) | 2 | 3 | 1
Chills (General disorders) | 5 | 10 | 1
Fatigue (General disorders) | 15 | 39 | 3
Influenza like illness (General disorders) | 1 | 3 | 0
Infusion site pain (General disorders) | 1 | 0 | 0
Injection site extravasation (General disorders) | 1 | 0 | 0
Local swelling (General disorders) | 1 | 1 | 0
Malaise (General disorders) | 0 | 3 | 0
Mucosal dryness (General disorders) | 0 | 3 | 0
Mucosal inflammation (General disorders) | 1 | 11 | 1
Oedema peripheral (General disorders) | 7 | 27 | 1
Pain (General disorders) | 3 | 4 | 0
Pyrexia (General disorders) | 8 | 20 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 2 | 3 | 0
Candidiasis (Infections and infestations) | 2 | 5 | 0
Cellulitis (Infections and infestations) | 3 | 5 | 0
Folliculitis (Infections and infestations) | 1 | 1 | 0
Fungal infection (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 1
Localised infection (Infections and infestations) | 0 | 1 | 1
Oral candidiasis (Infections and infestations) | 1 | 2 | 0
Pneumonia (Infections and infestations) | 1 | 2 | 0
Rash pustular (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 3 | 4 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 4 | 0
Urinary tract infection (Infections and infestations) | 1 | 7 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 2 | 0
Incision site complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Medical device pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Nail avulsion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 3 | 0
Procedural site reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Stent occlusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 6 | 4 | 0
Aspartate aminotransferase increased (Investigations) | 5 | 3 | 0
Blood albumin decreased (Investigations) | 1 | 3 | 0
Blood alkaline phosphatase increased (Investigations) | 4 | 1 | 0
Blood creatinine increased (Investigations) | 2 | 2 | 0
Blood urine present (Investigations) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 9 | 0
Platelet count decreased (Investigations) | 1 | 1 | 1
Weight decreased (Investigations) | 2 | 8 | 1
Weight increased (Investigations) | 1 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 9 | 22 | 2
Dehydration (Metabolism and nutrition disorders) | 6 | 12 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 4 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 4 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 3 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 12 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 4 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 4 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 10 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 5 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1
Bunion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Joint contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 10 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 9 | 0
Balance disorder (Nervous system disorders) | 2 | 3 | 0
Burning sensation (Nervous system disorders) | 2 | 2 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 8 | 13 | 2
Dysarthria (Nervous system disorders) | 1 | 1 | 0
Dysgeusia (Nervous system disorders) | 3 | 16 | 2
Head discomfort (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 7 | 9 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 4 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 5 | 29 | 2
Paraesthesia (Nervous system disorders) | 1 | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 3 | 0
Peripheral nerve palsy (Nervous system disorders) | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 3 | 0
Sinus headache (Nervous system disorders) | 1 | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 2 | 1
Agitation (Psychiatric disorders) | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 2 | 13 | 0
Confusional state (Psychiatric disorders) | 2 | 2 | 0
Depressed mood (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 8 | 0
Insomnia (Psychiatric disorders) | 7 | 13 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 0
Bladder spasm (Renal and urinary disorders) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 3 | 0
Haematuria (Renal and urinary disorders) | 1 | 1 | 0
Incontinence (Renal and urinary disorders) | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 2 | 0
Renal pain (Renal and urinary disorders) | 1 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0
Urinary tract disorder (Renal and urinary disorders) | 1 | 1 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 13 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 11 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 10 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 6 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 15 | 35 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 3 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 10 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 5 | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 2 | 2 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 4 | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 10 | 0
Rash (Skin and subcutaneous tissue disorders) | 7 | 22 | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Biliary drainage (Surgical and medical procedures) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 5 | 0
Flushing (Vascular disorders) | 2 | 2 | 0
Hypertension (Vascular disorders) | 1 | 3 | 0
Hypotension (Vascular disorders) | 3 | 5 | 0
Orthostatic hypotension (Vascular disorders) | 2 | 6 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution may publish the results of its findings if a multicenter publication is not forthcoming within 18 months after study completion. Institution shall provide Celgene with a copy of the papers prior to their submission; Celgene shall complete its review within 30 days after receipt. Upon Celgene's request, proposed publication or presentation can be delayed up to 60 additional days to enable Celgene to secure adequate intellectual property protection of patentable material.